CLINICAL TRIAL: NCT00298389
Title: Macrophage Phagocytosis in Chronic Obstructive Pulmonary Disease
Brief Title: Macrophage Phagocytosis in COPD
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 05/Q0404/111
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema; Chronic Bronchitis
Keywords: macrophage; phagocytosis; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non smokers: Non smokers included no history of respiratory or allergic disease, normal baseline spirometry
- Smokers: Smoking history of at least 10 pack years
- COPD: Patients with stable COPD

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) that have frequent chest infections are the patients most likely to become worse over time. Why these people are more susceptible to chest infections is not known. One reason might be that the white cells in their lungs called macrophages do not work properly. Normally, these cells remove all the debris inhaled into the lung. This can also include bacteria. In patients with COPD, these macrophages are not able to remove these particles. The research question addresses why this happens

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) comprises chronic bronchitis, small airways disease and emphysema. The major risk factor for the development of COPD is cigarette smoking therefore, the prevalence of this disease is increasing. COPD accounts for increasing numbers of hospital admissions due to increased numbers of chest infections and exacerbations. This may be related to the reduced capacity of macrophages from COPD patients to phagocytose bacteria and apoptotic cells. The reasons for this defect in the innate immune response in these subjects is unclear but there are suggestions that scavenger receptors may be altered by oxidative stress and reduce the phagocytotic pathway. This would be relevant in COPD, as increased oxidative stress is associated with cigarette smoking. We have preliminary data that shows a similar reduce phagocytotic response in monocyte-derived macrophages (MDM) from COPD patients compared with smokers and non-smokers. As these cells have not been exposed to oxidative stress other mechanisms may play a role in reducing phagocytosis. Using this MDM model, by taking blood from patients with COPD, we aim to investigate the mechanism of defective phagocytosis in COPD. We will measure the expression and regulation of cell surface scavenger receptors in cells of disease patients and control subjects and examine the signalling pathways leading to actin polymerization and phagosome formation. Finally, we aim to identify novel therapeutic strategies to reverse this effect and augment phagocytosis of macrophages in patients with COPD. Such a strategy would reduce chest infections and exacerbations and hence improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

Healthy non-smoking subjects:

All normal volunteers will meet the following criteria:

Age 21-75 years. No history of respiratory or allergic disease. Normal baseline spirometry as predicted for age, sex and height. Non-smokers. No history of upper respiratory tract infection in the preceding six weeks. Not taking regular medication

COPD subjects:

COPD is diagnosed according to American Thoracic Society, European Respiratory Society and British Thoracic Society guidelines by the doctors in Professor Barnes' COPD clinic.

All COPD volunteers will meet the following criteria:

Age between 35-75 years. A smoking history of at least 10 pack years. ( 1 pack year = 20 cigarettes per day for 1 year) FEV1:FVC ratio of <0.7, post-bronchodilator FEV1 of <85% predicted, reversibility with inhaled beta2-agonist of <15% of predicted FEV1: all three criteria are required.

Exclusion Criteria:

Subjects will not included in this study if they meet any of the following exclusion criteria:

Clinically significant findings in the medical history or on physical examination other than those of COPD in the COPD group.

Pregnant women or mothers who are breastfeeding. Subjects who are unable to give informed consent.-

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, smokers without COPD and COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise E Donnelly, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taylor AE, Finney-Hayward TK, Quint JK, Thomas CM, Tudhope SJ, Wedzicha JA, Barnes PJ, Donnelly LE. Defective macrophage phagocytosis of bacteria in COPD. Eur Respir J. 2010 May;35(5):1039-47. doi: 10.1183/09031936.00036709. Epub 2009 Nov 6. PMID 19897561

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non Smokers | Smokers | COPD
Started | 20 | 17 | 19
Completed | 20 | 17 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non Smokers | Smokers | COPD | Total
Number analyzed (Participants) | 20 | 17 | 19 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (3) | 53 (2) | 70 (2) | 57 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 24
  Male | 11 | 10 | 11 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 17 | 19 | 56
Smoking history [Mean (Standard Deviation); unit: pack/years] | 0 (0) | 33 (4.6) | 45 (4.9) | 15.3 (20)
FEV1 (%predicted) [Mean (Standard Deviation); unit: percent predicted] | 102.7 (2.6) | 93.8 (3.8) | 50.6 (4.0) | 80.5 (20)

OUTCOME MEASURES:

1. Primary Outcome: Phagocytosis of H. Influenzae Concentration
Description: Measurement of phagocytosis in vitro, Phagocytosis of H. influenzae concentration
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: relative fluorescence unit
Arm/Group | Non Smokers | Smokers | COPD
Number analyzed (Participants) | 20 | 17 | 19
relative fluorescence unit
  concentration 0.3g/ml | 0.042 (0.008) | 0.042 (0.007) | 0.014 (0.002)
  concentration 1g/ml | 0.06 (0.01) | 0.059 (0.008) | 0.025 (0.004)
Statistical Analysis 1: Comparison: Non Smokers vs Smokers vs COPD; Test type: Superiority; p = 0.05, Kruskal-Wallis — calculated

2. Primary Outcome: Phagocytosis of S. Pneumoniae Concentration
Description: Measurement of phagocytosis in vitro, Phagocytosis of S. pneumoniae concentration
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: relative fluescence
Arm/Group | Non Smokers | Smokers | COPD
Number analyzed (Participants) | 20 | 17 | 19
relative fluescence
  concentration 0.3g/ml | 0.066 (0.02) | 0.056 (0.012) | 0.012 (0.011)
  concentration 1g/ml | 0.077 (0.021) | 0.072 (0.016) | 0.022 (0.014)
Statistical Analysis 1: Comparison: Non Smokers vs Smokers vs COPD; Test type: Superiority; p = 0.05, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Non Smokers | Smokers | COPD
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes